CLINICAL TRIAL: NCT03904511
Title: Safety, Tolerability and Behavioural Effects of Souroubea-Platanus in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Souroubea Botanicals Inc. (Unknown)
Responsible Party: Principal Investigator, Jakov Shlik, Clinical Director, OSI Clinic at The Royal, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018005
Record Dates: First submitted 2019-03-16; First posted 2019-04-05 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Anxiety; Stress, Psychological
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose Souroubea-Platanus (Experimental): 190 mg souroubea-platanus preparation in vegicap. Administered once daily for 14 days.
  Interventions: Other: Souroubea-Platanus Preparation
- High Dose Souroubea-Platanus (Experimental): 380 mg souroubea-platanus preparation in vegicap. Administered once daily for 14 days.
  Interventions: Other: Souroubea-Platanus Preparation
- Placebo (Placebo Comparator): Inert placebo in an identical vegicap to the experimental treatment groups. Administered once daily for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Souroubea-Platanus Preparation — Extracts of S. Sympetala and P. occidentalis.
  Arms: High Dose Souroubea-Platanus; Low Dose Souroubea-Platanus
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Souroubea sympetala extracts have shown anxiolytic properties in animal models. Souroubea and its active principle betulinic acid appear to exert these effects by acting as an agonist for the benzodiazepine (BZD) binding site of the GABAA receptor with no withdrawal effects on food intake, locomotor activity, or other symptoms typically associated with BZD agonism. As such, this may offer a valuable source for an alternative anti-anxiety treatment.

The primary objective of this study is to (1) to evaluate the safety and tolerability of a single daily dose of an extract of a mixture of Souroubea spp. leaf and small branch material and Platanus spp. bark when administered orally over two weeks in healthy volunteers. Based on its safety in canine trials, we hypothesize that Souroubea-Platanus (SP) preparation will be well tolerated with adverse event profile similar to placebo.

The secondary objective is (2) to establish whether some of the anxiolytic properties of Souroubea-platanus seen in animal models will translate to human participants. We hypothesize that Souroubea-Platanus preparation will demonstrate anxiolytic and/or stress-reduction properties as indicated by salivary cortisol levels and self-report measures of anxiety.

DETAILED DESCRIPTION:
Background

Within Latin American indigenous communities tea brewed from fresh or dried crushed Souroubea leaves is used to treat Susto, a culture-bound syndrome resembling manifestations of Anxiety Disorders. Souroubea sympetala (Ss) leaf extract has shown to be effective as an anxiolytic in animal models, and betulinic acid (BA) is one of the active molecules responsible for mediating this effect.

Plant-based natural products are sought by many individuals as alternatives or supplements to standard medical care. As a result, more research is required in order to develop botanical treatments that are evidence-based, safe and guided by health practitioners. Souroubea-Platanus may offer such alternative.

Safety

Evidence suggests that Souroubea-Platanus was well tolerated in Beagles in a 28-day pilot study at 8x recommended dose, producing significant reductions in plasma cortisol 1h post-administration without any adverse reactions, except slightly reduced platelet count in 2 animals attributed to infection with Ehrlichia canis, likely contracted prior to the study onset. In a follow-up 16 beagles and up to 5x the recommended does for 28 days such decrease in platelet count was not observed, no there were any other adverse events. No adverse events have been reported in animals for the animal health product version of the drug (Zentrol) that has been on the market for 2 years. The naturalistic observations of Souroubea consumption suggest that it is safe for human use, however, this has not been established in a formal study. In addition, drug interactions have occurred with some herbal products, particularly those that strongly inhibit or induce CYP enzymes. As Souroubea may act on the BDZ binding site of the GABAA receptor, possible side-effects and symptoms similar to those associated with benzodiazepine anxiolytics are possible.

Clinical Relevance

The study has significant clinical relevance for anxiety and stress-related disorders and may lead to developing a new anxiolytic agent or supplement with more selective effects and reduced risks for the patients.

Overview of study design

Forty-five healthy adult volunteers will be enrolled in the single-center, randomized, double-blind, parallel group study. Power analysis revealed that to achieve a power of 0.80, with an estimated effect size of 0.40 (estimate based on rodent studies), a total sample size of 42 would be required. Accounting for approximately 10% predicted participant dropout rate per group, it is expected that 45 participants will be enrolled in the study.

Participants will be randomly assigned to one of the 3 treatment groups with 15 individuals in each for detecting a dose-response effect. Treatment groups will be either (a) 190mg extract (b) 380mg extract, or (c) inert placebo, all in identical vegicaps.

Capsules containing the placebo and the extracts will be produced under GMP conditions. In accordance with Health Canada guidelines, extract will conform to the acceptable limits for heavy metal and biological contamination. The placebo will consist of microcrystalline cellulose suitable for use in foods.

The capsules will be taken once a day in the morning with water for 2 consecutive weeks. The safety evaluations will be conducted at screening and repeated at the end of the 2-week study period. Adverse events will be evaluated after 1 week and 2 weeks of treatment and 1 week after discontinuation. The participants will be asked to maintain their regular lifestyle and diet during the study period so long as those habits do not violate the study exclusion criteria.

Participants will be asked to take the capsules at the same time every morning. Compliance will be facilitated by daily reminders by e-mail, text, or phone call and a review of the returned medication vials.

The participants will have 24-hour phone access to the study physician for emergencies.

Participant Compensation

Participants will be reimbursed for their time in participation, as well as for transportation and parking costs on prorated basis corresponding to minimal hourly wage.

Randomization and blinding

Blinded treatment will be used to reduce potential bias during data collection and evaluation of clinical endpoints. Participant numbers will be assigned in sequential order as participants enroll in the study. All participants will be asked to come in at the same time for all testing periods after screening (Days 1, 7, 14, and 21) in order to account for time-of-day effects on cortisol.

Participants will be assigned to one of the treatment groups according to a computer generated randomization schedule prepared by contracted pharmacy personnel. The randomization will be balanced by using permuted blocks. Pharmacy personnel will package and label study drug for each participant.

The study investigator or his/her designate and study participant will remain blind to the participants' group until the completion of the study. The blind should be broken only if in emergency requiring knowing the treatment status of the participant.

Study procedures

1. Baseline screening will include:

   1. Medical history, physical examination, and vital signs, including temperature, heart rate, respiratory rate and blood pressure;
   2. Mental status examination, including completion of the DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure - Adult with follow-up on any items rated as present in at least mild degree;
   3. Laboratory tests and urine drug screen as described below;
   4. Serum pregnancy test for females of childbearing potential; must not be pregnant
2. Safety evaluations:

   1. Each volunteer will provide a blood and urine sample in the morning, within 14 days before the start of the study (baseline), 7 days after the first dose, and on the last day of the study (day 14). Body weight will be measured at baseline and day 14. Physical examination including vital signs and inquiry of adverse events will be performed on days 7 and 14. Additional evaluation of adverse events will be done one week after discontinuation of the study drug. Vital signs will be monitored until 1 hour after administration of the first dose.

The following laboratory parameters will be measured:

* complete blood count: white blood cell (WBC) count with differential, red blood cell (RBC) count, hemoglobin, hematocrit and indices, platelet count;
* chemistry panel: glucose, calcium, electrolytes (sodium, potassium, chloride), BUN, creatinine, albumin, total protein, alkaline phosphatase, gamma glutamyl transferase, aspartate aminotransferase, alanine aminotransferase, bilirubin, creatine kinase;
* urinalysis will be standard, microscopic if indicated;
* salivary cortisol will be measured as a stress indicator.

Pregnancy testing in females will consist of a serum test (for convenience, since other blood samples are already being collected during screening; this should not normally require additional venipuncture).

Saliva samples will be collected using sterile saliva sample tubes. Blood and urine samples will be collected at the clinical laboratory. Blood samples will be drawn by venipuncture.

Records of health data identifying participants will be kept on record for 25 years before being destroyed; all records will be kept confidential during that time.

Behavioural evaluations

1. State-Trait Anxiety Inventory (STAI) on Days 1 (baseline and 1 hour post-dose), 7 and 14.
2. DSM-5 Self-rated Level 2 anxiety adult short form on Days 1, 7, and 14
3. Cortisol (physiological marker of stress): salivary concentration; analysis - difference between pre- and 1 h post dose on Day 1, max changes from baseline and group x time effects and interactions.

Data analysis

Statistical means and standard deviations will be calculated for each continuous variable. ANOVA followed by post hoc Tukey's test will be used to evaluate significant differences among dose groups and different days. A P-value of 0.05 will be considered as the level of significant difference in the analysis of the data. Behavioural variables will be analyzed using mixed effects ANOVA for repeated measures where appropriate.

Transformations for non-normality and/or corrective procedures will be applied if data is found to be non-normally distributed or otherwise in violation of the assumptions of the statistical tests.

STAI: the total sum scores (T-scores); analysis - max changes from baseline and group x time effects and interactions.

Cortisol: salivary concentration; analysis - difference between pre- and 1 h post dose on Day 1, max changes from baseline and group x time effects and interactions.

Safety evaluations will be based on the baseline to treatment-period differences in laboratory tests, physical examinations, vital signs and the incidence of adverse events.

Adverse events reporting

All adverse events (AE) regardless of casual relationship with investigational treatment will be recorded. An AE will be considered treatment-emergent if it is new in onset or aggravated in severity or frequency following administration of the investigational agent. All treatment emergent AE will be followed until resolution or a stable clinical endpoint.

Serious AE, e.g. any AE that is fatal, immediately life threatening, requires or prolongs hospitalization, causes permanent or significant disability will be reported to Health Canada and IRB and immediately addressed medically as appropriate.

Participants will be encouraged to report AEs spontaneously or in response to general, non-directed questioning. All treatment-emergent AEs will be recorded in the source document using medical terminology.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18-70 years
2. Females of childbearing potential must use reliable contraception during the study period; acceptable methods of birth control include all hormonal methods, IUDs, complete abstinence, effective physical barriers (e.g. condoms), or confirmed vasectomy of partner (if that information is volunteered by the participant)
3. Participants must be in good health status based on medical history and physical examination, including vital signs and clinical laboratory tests
4. Participants must refrain from taking any prescription or over the counter medication within the 14 days prior to the beginning of the study and during the study period
5. Participants must be non-smokers or light/occasional smokers (not more than 10 cigarettes per day)
6. Alcohol consumption should not exceed 3 drinks on any single day and no more than 7 drinks per week in women and no more than 4 drinks on any single day and no more than 14 drinks per week for men
7. BMI of 18.5-30 kg/m2 excluding markedly underweight and obese individuals
8. Participants must be willing to give written informed consent after the nature of the study has been fully explained

Exclusion Criteria:

1. Participants demonstrating uncontrolled clinically significant physical disease or abnormal laboratory test results within 14 days prior to the start of the study
2. Participants with current or history of alcohol or drug use disorder
3. Participants with any history of significant drug super-sensitivity, anaphylaxis, or anaphylactic reaction
4. Participants taking prescription medication or OTC medication within 14 days prior to inclusion
5. Participants who have a history of any significant psychiatric disorder or currently significant psychiatric symptoms
6. Participants with a family history of serious mental illness in first-degree relatives
7. Participants in a situation or having any condition which, in the opinion of the investigator, may interfere with optimal participation in the study
8. Participants testing positive for amphetamine, cannabinoids, cocaine, barbiturates, benzodiazepines, opioids or hallucinogens
9. Use of other non-prescription natural health products with known anti-anxiety effects
10. Known allergy to any of the medicinal and non-medicinal ingredients in any conditions of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Weight | Change from baseline weight (screening) in kg until day 14 of the protocol.
  Participant weight (kilograms)
Heart rate | Change from baseline (screening) bpm until day 14 of the protocol.
  Heart rate (bpm)
Blood pressure | Change from baseline (screening) blood pressure until day 14 of the protocol.
  Systolic and Diastolic Blood pressure (mmhg)
Body temperature | Change from baseline (screening) body temperature in degrees Fahrenheit until day 14 of the protocol.
  Body temperature (degrees Fahrenheit).
White blood cell (WBC) count (per L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  White blood cell (WBC) count (per L)
Red blood cell (RBC) count (per L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Red blood cell (RBC) count (per L)
Hemoglobin (g/L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Hemoglobin (g/L)
Hematocrit (vol%) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Hematocrit (vol%)
Platelet count (per L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Platelet count (per L)
Blood Glucose (mg/dL) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Blood Glucose (mg/dL)
Serum calcium (mg/dL) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum calcium (mg/dL)
Serum potassium (mEq/L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum potassium (mEq/L)
Serum sodium (mEq/L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum sodium (mEq/L)
Serum chloride (mEq/L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum chloride (mEq/L)
BUN; blood urea nitrogen (mg/dL) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  BUN; blood urea nitrogen (mg/dL)
Creatinine (mg/dL) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Creatinine (mg/dL)
Serum albumin (g/dL) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum albumin (g/dL)
Serum total protein (g/dL) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum total protein (g/dL)
Serum ALP; Alkaline phosphatase (U/L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum ALP; Alkaline phosphatase (U/L)
Serum GGT; Gamma glutamyl transferase (U/L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum GGT; Gamma glutamyl transferase (U/L)
Serum AST; Aspartate aminotransferase (U/L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum AST; Aspartate aminotransferase (U/L)
Serum ALT ; Alanine aminotransferase (U/L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum ALT ; Alanine aminotransferase (U/L)
Serum CK; Creatinine Kinase (U/L) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum CK; Creatinine Kinase (U/L)
Serum Bilirubin (mg/dL) | Change from baseline (screening) in any parameters until day 14 of the protocol.
  Serum Bilirubin (mg/dL)
Urinary Glucose (mmol/L) | Change from baseline (screening) until day 14 of the protocol.
  Urinary Glucose (mmol/L)
Urinary ketones (mg/dL) | Change from baseline (screening) until day 14 of the protocol.
  Urinary ketones (mg/dL)
Urinary protein (mg/dL) | Change from baseline (screening) until day 14 of the protocol.
  Urinary protein (mg/dL)
Urinalysis; visual inspection | Change from baseline (screening) until day 14 of the protocol.
  Urinalysis; visual inspection, and microscopic visual examination if abnormal results present during visual inspection or on any of the chemistry panels.
Urinary pH | Change from baseline (screening) until day 14 of the protocol.
  Urinary pH
Urinary leukocytes (U/L) | Change from baseline (screening) until day 14 of the protocol.
  Urinary leukocytes (U/L)
UBG; Urobilinogen (mg/dL) | Change from baseline (screening) until day 14 of the protocol.
  UBG; Urobilinogen (mg/dL)
Urinary nitrites | Change from baseline (screening) until day 14 of the protocol.
  Urinary nitrites
Urinary specific gravity (S.G.) | Change from baseline (screening) until day 14 of the protocol.
  Urinary specific gravity (S.G.)

SECONDARY OUTCOMES:
DSM-5 Self-rated Level 2 Anxiety | DSM-5 Self-rated Level 2 Anxiety to be completed on days 1, 7, and 14 of the 21-day protocol.
  The DSM-5 Level 2 Anxiety Adult measure has 7 items that assesses the domain of anxiety in individuals age 18 and older. All items are rated on a 5-point scale. Higher scores indicate greater anxiety. The DSM-5 Self-rated Level 2 Anxiety has a minimum score of 7 and a maximum score of 35.
State-Trait Anxiety Inventory for Adults (STAI-AD) | Change from baseline until day 21 of the protocol.
  The State-Trait Anxiety Inventory (STAI) has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale. Higher scores indicate greater anxiety. The STAI has a score range of 20-80, with a minimum score of 20 and a maximum score of 80.
Concentration of cortisol in saliva, measured in ng/sample | Change from baseline unil day 21 of the protocol.
  Concentration of cortisol in saliva, measured in ng/sample

CONTACTS AND LOCATIONS:
Overall Officials: Jakov Shlik, MD, Principal Investigator — University of Ottawa
Locations (1):
- The Royal's Institute of Mental Health Research (IMHR) affiliated with the University of Ottawa, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Bourbonnais-Spear N, Awad R, Merali Z, Maquin P, Cal V, Arnason JT. Ethnopharmacological investigation of plants used to treat susto, a folk illness. J Ethnopharmacol. 2007 Feb 12;109(3):380-7. doi: 10.1016/j.jep.2006.08.004. Epub 2006 Sep 10. PMID 17071033
- [Background] Crandon L. Why susto. Ethnology 1983;22:153-167.
- [Background] Klein J. Susto: the anthropological study of diseases of adaptation. Soc Sci Med (1967). 1978 Jan;12(1B):23-8. No abstract available. PMID 644342
- [Background] Rubel AJ. The epidemiology of a folk illness: Susto in Hispanic America. Ethnology 1964;3:268-283.
- [Background] Signorini I. Patterns of fright: multiple concepts of susto in a Nahua-Ladino Community of the Sierra de Puebla (Mexico). Ethnology 1982;21:313-323.
- [Background] Bourbonnais-Spear N. Ethnobotany and ethnopharmacology of Q'eqchi'Maya medicinal plants from southern Belize used for ethnopsychiatric and neurological purposes. University of Ottawa (Canada), 2005.
- [Background] Puniani E, Cayer C, Kent P, Mullally M, Sanchez-Vindas P, Poveda Alvarez L, Cal V, Merali Z, Arnason JT, Durst T. Ethnopharmacology of Souroubea sympetala and Souroubea gilgii (Marcgraviaceae) and identification of betulinic acid as an anxiolytic principle. Phytochemistry. 2015 May;113:73-8. doi: 10.1016/j.phytochem.2014.02.017. Epub 2014 Mar 15. PMID 24641939
- [Background] Mullally M, Mimeault C, Rojas MO, Vindas PS, Garcia M, Alvarez LP, et al. A botanical extract of Souroubea sympetala and its active principle, betulinic acid, attenuate the cortisol response to a stressor in rainbow trout, Oncorhynchus mykiss. Aquaculture 2017;468:26-31.
- [Background] Mullally M, Cayer C, Kramp K, Otarola Rojas M, Sanchez Vindas P, Garcia M, Poveda Alvarez L, Durst T, Merali Z, Trudeau VL, Arnason JT. Souroubea sympetala (Marcgraviaceae): a medicinal plant that exerts anxiolysis through interaction with the GABAA benzodiazepine receptor. Can J Physiol Pharmacol. 2014 Sep;92(9):758-64. doi: 10.1139/cjpp-2014-0213. Epub 2014 Jul 28. PMID 25140794
- [Background] Cayer C. In vivo behavioural characterization of anxiolytic botanicals: Souroubea sympetala. PhD Thesis. Masters Thesis submitted to the University of Ottawa, 2011.
- [Background] Kessler RC, Soukup J, Davis RB, Foster DF, Wilkey SA, Van Rompay MI, Eisenberg DM. The use of complementary and alternative therapies to treat anxiety and depression in the United States. Am J Psychiatry. 2001 Feb;158(2):289-94. doi: 10.1176/appi.ajp.158.2.289. PMID 11156813
- [Background] Villalobos P, Baker J, Sanchez Vindas P, Durst T, Masic A, Arnason JT. Clinical Observations and Safety Profile of Oral Herbal Products, Souroubea and Platanus Spp; a Pilot-Toxicology Study in Dogs. Acta Vet (Beogr) 2014;64:269-275.
- [Background] Masic A, Liu R, Simkus K, Wilson J, Baker J, Sanchez P, Saleem A, Harris CC, Durst T, Arnason JT. Safety evaluation of a new anxiolytic product containing botanicals Souroubea spp. and Platanus spp. in dogs. Can J Vet Res. 2018 Jan;82(1):3-11. PMID 29382964
- [Background] Liu R, Ahmed F, Cayer C, Mullally M, Carballo AF, Rojas MO, Garcia M, Baker J, Masic A, Sanchez PE, Poveda L, Merali Z, Durst T, Arnason JT. New Botanical Anxiolytics for Use in Companion Animals and Humans. AAPS J. 2017 Nov;19(6):1626-1631. doi: 10.1208/s12248-017-0144-y. Epub 2017 Sep 11. PMID 28895076
- [Background] Smith RD, Ristic M, Huxsoll DL, Baylor RA. Platelet kinetics in canine ehrlichiosis: evidence for increased platelet destruction as the cause of thrombocytopenia. Infect Immun. 1975 Jun;11(6):1216-21. doi: 10.1128/iai.11.6.1216-1221.1975. PMID 1140846
- [Background] Romero LE, Meneses AI, Salazar L, Jimenez M, Romero JJ, Aguiar DM, Labruna MB, Dolz G. First isolation and molecular characterization of Ehrlichia canis in Costa Rica, Central America. Res Vet Sci. 2011 Aug;91(1):95-97. doi: 10.1016/j.rvsc.2010.07.021. Epub 2010 Aug 17. PMID 20723954
- [Background] Miller NS, Gold MS. Benzodiazepines: a major problem. Introduction. J Subst Abuse Treat. 1991;8(1-2):3-7. doi: 10.1016/0740-5472(91)90021-2. PMID 1675690
- [Background] Mullally M, Kramp K, Cayer C, Saleem A, Ahmed F, McRae C, Baker J, Goulah A, Otorola M, Sanchez P, Garcia M, Poveda L, Merali Z, Durst T, Trudeau VL, Arnason JT. Anxiolytic activity of a supercritical carbon dioxide extract of Souroubea sympetala (Marcgraviaceae). Phytother Res. 2011 Feb;25(2):264-70. doi: 10.1002/ptr.3246. PMID 20648677